CLINICAL TRIAL: NCT04864080
Title: Transdiagnostic Cognitive Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEUR-2020-29420
Record Dates: First submitted 2021-01-20; First posted 2021-04-28 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pain; Depression
MeSH Terms: conditions — Pain; Depression | interventions — Patient Health Questionnaire

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Comparison Group (Active Comparator): Behavioral tasks and surveys online.
  Interventions: Behavioral: Computer game/task; Behavioral: Health surveys online
- Pain/Depression patients from clinic (Experimental): MRI, TMS and EEG, and behavioral tasks and surveys online.
  Interventions: Behavioral: Computer game/task; Behavioral: Health surveys online

INTERVENTIONS:
Behavioral: Computer game/task — N-back, COGED, PacMan game, Bandit task, Websurf task.
  Other Names: Behavioral tasks online and in-person.
Behavioral: Health surveys online — Health surveys to study themes like pain, sleep, depression and anxiety, and PTSD.
  Other Names: PHQ-9, MASQ, GAD-7

SUMMARY:
The overall objective of this study is to determine the feasibility of identifying transdiagnostic biomarkers of cognitive function mediated by neuromodulation of the dorsolateral prefrontal cortex that are translatable across disease groups in order to more accurately phenotype clusters of cognitive dysfunction. Completing behavioral paradigms with electrophysiology and TMS is a challenging frontier. This study focuses on the feasibility of such an endeavor for those with chronic pain or depression as well as healthy controls.

DETAILED DESCRIPTION:
This study aims to test the feasibility of procedures aimed at discovering transdiagnostic biomarkers for cognitive impairment in chronic pain and depression. Fifteen healthy control participants and 15 participants from each disease group (chronic pain, depression) will be recruited.

Using a task-based fmri, TMS will be targeted for priming of the Left DLPFC. EEG will be used during our behavioral paradigm to compare changes in DLPFC function before and after primed TMS.

ELIGIBILITY:
Arm 1, healthy controls:

Inclusion Criteria:

* Have access to the online study platform.

Exclusion Criteria:

* under 18, non-English speaking

Arm 2: pain and depression:

Inclusion Criteria:

* Pain or depression

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility for all aspects of the study | 1-7 days
  Feasibility; the overall objective of this study is to determine the feasibility of identifying transdiagnostic biomarkers of cognitive function mediated by neuromodulation of the dorsolateral prefrontal cortex that are translatable across disease groups in order to more accurately phenotype clusters of cognitive dysfunction. Completing behavioral paradigms with electrophysiology and TMS is a challenging frontier. This study focuses on the feasibility of such an endeavor for those with chronic pain or depression as well as healthy controls.

SECONDARY OUTCOMES:
Acceptability | 1-7 days
  Sum total of acceptability rating scale of study procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Chung SW, Rogasch NC, Hoy KE, Fitzgerald PB. The effect of single and repeated prefrontal intermittent theta burst stimulation on cortical reactivity and working memory. Brain Stimul. 2018 May-Jun;11(3):566-574. doi: 10.1016/j.brs.2018.01.002. Epub 2018 Jan 8. PMID 29352668
- [Background] Schicktanz N, Fastenrath M, Milnik A, Spalek K, Auschra B, Nyffeler T, Papassotiropoulos A, de Quervain DJ, Schwegler K. Continuous theta burst stimulation over the left dorsolateral prefrontal cortex decreases medium load working memory performance in healthy humans. PLoS One. 2015 Mar 17;10(3):e0120640. doi: 10.1371/journal.pone.0120640. eCollection 2015. PMID 25781012
- [Background] Vekony T, Nemeth VL, Holczer A, Kocsis K, Kincses ZT, Vecsei L, Must A. Continuous theta-burst stimulation over the dorsolateral prefrontal cortex inhibits improvement on a working memory task. Sci Rep. 2018 Oct 4;8(1):14835. doi: 10.1038/s41598-018-33187-3. PMID 30287868
- [Background] Ekhtiari H, Tavakoli H, Addolorato G, Baeken C, Bonci A, Campanella S, Castelo-Branco L, Challet-Bouju G, Clark VP, Claus E, Dannon PN, Del Felice A, den Uyl T, Diana M, di Giannantonio M, Fedota JR, Fitzgerald P, Gallimberti L, Grall-Bronnec M, Herremans SC, Herrmann MJ, Jamil A, Khedr E, Kouimtsidis C, Kozak K, Krupitsky E, Lamm C, Lechner WV, Madeo G, Malmir N, Martinotti G, McDonald WM, Montemitro C, Nakamura-Palacios EM, Nasehi M, Noel X, Nosratabadi M, Paulus M, Pettorruso M, Pradhan B, Praharaj SK, Rafferty H, Sahlem G, Salmeron BJ, Sauvaget A, Schluter RS, Sergiou C, Shahbabaie A, Sheffer C, Spagnolo PA, Steele VR, Yuan TF, van Dongen JDM, Van Waes V, Venkatasubramanian G, Verdejo-Garcia A, Verveer I, Welsh JW, Wesley MJ, Witkiewitz K, Yavari F, Zarrindast MR, Zawertailo L, Zhang X, Cha YH, George TP, Frohlich F, Goudriaan AE, Fecteau S, Daughters SB, Stein EA, Fregni F, Nitsche MA, Zangen A, Bikson M, Hanlon CA. Transcranial electrical and magnetic stimulation (tES and TMS) for addiction medicine: A consensus paper on the present state of the science and the road ahead. Neurosci Biobehav Rev. 2019 Sep;104:118-140. doi: 10.1016/j.neubiorev.2019.06.007. Epub 2019 Jul 2. PMID 31271802
- [Background] McNeill A, Monk RL, Qureshi AW, Makris S, Heim D. Continuous Theta Burst Transcranial Magnetic Stimulation of the Right Dorsolateral Prefrontal Cortex Impairs Inhibitory Control and Increases Alcohol Consumption. Cogn Affect Behav Neurosci. 2018 Dec;18(6):1198-1206. doi: 10.3758/s13415-018-0631-3. PMID 30132267
- [Background] Boggio PS, Ferrucci R, Rigonatti SP, Covre P, Nitsche M, Pascual-Leone A, Fregni F. Effects of transcranial direct current stimulation on working memory in patients with Parkinson's disease. J Neurol Sci. 2006 Nov 1;249(1):31-8. doi: 10.1016/j.jns.2006.05.062. Epub 2006 Jul 14. PMID 16843494
- [Background] Short BE, Borckardt JJ, Anderson BS, Frohman H, Beam W, Reeves ST, George MS. Ten sessions of adjunctive left prefrontal rTMS significantly reduces fibromyalgia pain: a randomized, controlled pilot study. Pain. 2011 Nov;152(11):2477-2484. doi: 10.1016/j.pain.2011.05.033. Epub 2011 Jul 20. PMID 21764215
- [Background] To WT, De Ridder D, Hart J Jr, Vanneste S. Changing Brain Networks Through Non-invasive Neuromodulation. Front Hum Neurosci. 2018 Apr 13;12:128. doi: 10.3389/fnhum.2018.00128. eCollection 2018. PMID 29706876
- [Background] Zilverstand A, Huang AS, Alia-Klein N, Goldstein RZ. Neuroimaging Impaired Response Inhibition and Salience Attribution in Human Drug Addiction: A Systematic Review. Neuron. 2018 Jun 6;98(5):886-903. doi: 10.1016/j.neuron.2018.03.048. PMID 29879391
- [Background] Sheng J, Liu S, Wang Y, Cui R, Zhang X. The Link between Depression and Chronic Pain: Neural Mechanisms in the Brain. Neural Plast. 2017;2017:9724371. doi: 10.1155/2017/9724371. Epub 2017 Jun 19. PMID 28706741
- [Background] Moran TP, Jendrusina AA, Moser JS. The psychometric properties of the late positive potential during emotion processing and regulation. Brain Res. 2013 Jun 21;1516:66-75. doi: 10.1016/j.brainres.2013.04.018. Epub 2013 Apr 17. PMID 23603408